CLINICAL TRIAL: NCT00148824
Title: Immunological Efficacy of a Prime-Boost Strategy Combining a 7-Valent Pneumococcal Conjugate Vaccine (PCV) Followed by a 23-Valent Pneumococcal Polysaccharide Vaccine (PPV) Versus PPV Alone in HIV-Infected Adults. ANRS 114 PNEUMOVAC.
Brief Title: Antibody Responses to Pneumococcal Vaccines Among HIV-Infected Adults.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 114 PNEUMOVAC
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections
Keywords: HIV infections; Pneumococcal vaccines; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Vaccines

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugate vaccine (vaccine)
Biological: 23-valent pneumococcal conjugate vaccine (vaccine)

SUMMARY:
Streptococcus pneumoniae is the major cause of bacterial infection in HIV-infected patients. The current pneumococcal vaccine is poorly efficacious in patients with a CD4 cell count lower than 500/mm3. This study will test the efficacy and safety of a new pneumococcal vaccine strategy in patients with a CD4 cell count between 200 and 500/mm3.

DETAILED DESCRIPTION:
Streptococcus pneumoniae (SP) is the major cause of bacterial infection in HIV-infected patients. The 23-valent pneumococcal polysaccharide (PPV) is poorly immunogenic in patients with CD4 below 500 cells/mm3. The purpose of this multicentric national study is to evaluate whether a prime with a 7-valent pneumococcal conjugate vaccine (PCV), able to induce immunological memory, would improve immunogenicity against SP polysaccharides. 212 HIV-1 infected patients, with a CD4 count between 200 and 500/mm3, will be randomly assigned to one of two vaccine groups: PCV at Week 0 followed by PPV at Week 4 or PPV alone at Week 4. Evaluation will be done at week 8. The primary endpoint is the proportion of patients who had antibody responses against 7 pneumococcal polysaccharides at Week 8. Secondary endpoints include the persistence of antibody responses at Weeks 24 and 96, vaccines safety and occurrence of pneumococcal disease over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with proven HIV-1 infection
* Naïve or antiretroviral experienced
* CD4 cell count between 200 and 500/mm3
* Plasma HIV RNA load lower than 4 log10 copies/mL
* Signed written informed consent

Exclusion Criteria:

* Immunotherapy
* Immunization with the PPV within the past 5 years
* Splenectomy
* Use of intravenous immunoglobulin within the past 2 months
* Chemotherapy or radiation
* Any other vaccination within the past 2 months
* Severe renal failure
* End-stage liver disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212
Dates: Start 2003-02; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients responders to 7 pneumococcal polysaccharides at W8

SECONDARY OUTCOMES:
Persistence of antibody responses at W24 and W96
Clinical tolerance of pneumococcal vaccines at W8
Evolution of the CD4 count and plasma HIV RNA load
Immunological substudy (predictive factors of the antibody responses) at W24

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lesprit, MD, Principal Investigator — Service d'Immunologie Clinique, Créteil, 94010, France; Geneviève Chêne, MD, PhD, Study Director — INSERM unité 593

REFERENCES:
- [Derived] Rabian C, Tschope I, Lesprit P, Katlama C, Molina JM, Meynard JL, Delfraissy JF, Chene G, Levy Y; ANRS 114 Pneumovac Study Group. Cellular CD4 T cell responses to the diphtheria-derived carrier protein of conjugated pneumococcal vaccine and antibody response to pneumococcal vaccination in HIV-infected adults. Clin Infect Dis. 2010 Apr 15;50(8):1174-83. doi: 10.1086/651418. PMID 20210645